CLINICAL TRIAL: NCT02429817
Title: Tomographic Comparison of Aerosol Lung Distribution With Two Nebulizers Through a High Flow Nasal Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Aerospect-02
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Pulmonary aerosol distribution; SPECT-CT analysis; High flow nasal cannula; Vibrating-mesh nebulizer; Jet nebulizer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Aeroneb Solo (Active Comparator): Subjects inhaled radiolabelled aerosol via the Aeroneb Solo connected to the high flow nasal cannula.
  Interventions: Drug: Technetium-99m - Diethylenetriaminepentaacetic acid; Device: Aeroneb Solo; Other: Single photon emission computed tomography; Other: Spirometry
- Standard Jet Nebulizer (Active Comparator): Subjects inhaled radiolabelled aerosol via the jet nebulizer connected to the high flow nasal cannula.
  Interventions: Drug: Technetium-99m - Diethylenetriaminepentaacetic acid; Device: Jet Nebulizer; Other: Single photon emission computed tomography; Other: Spirometry

INTERVENTIONS:
Drug: Technetium-99m - Diethylenetriaminepentaacetic acid — 99mTc-DTPA solution placed on the nebulizer reservoir
Device: Aeroneb Solo
  Arms: Aeroneb Solo
Device: Jet Nebulizer
  Arms: Standard Jet Nebulizer
Other: Single photon emission computed tomography — Imaging technique to investigate lung aerosol distribution
Other: Spirometry — FEV1, FVC assessment

SUMMARY:
Vibrating-mesh nebulizers ensure currently the best deposition output and are recommended in routine use in intensive care unit. However, jet nebulizers remain the most frequently used nebulizers.

On a bench study, aerosol delivery through a high flow nasal cannula (HFNC) was increased using a vibrating-mesh nebulizer as compared to a jet nebulizer.

Lung distribution of nebulized particles delivered through a HFNC has never been investigated in vivo. The aim of this study was to compare aerosol lung distribution with both nebulizers through a HFNC by SPECT-CT.

ELIGIBILITY:
Inclusion Criteria:

* Healthy respiratory function

Exclusion Criteria:

* Pulmonary disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary deposition | Immediately after nebulization by imaging technique, expected average of 15 minutes
  Single photon emission tomography combined with a CT-scan

SECONDARY OUTCOMES:
Three-dimensional penetration index | immediately after the nebulization by imaging assessment, expected average of 30 minutes

OTHER OUTCOMES:
Spirometry | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium